CLINICAL TRIAL: NCT04669249
Title: PROCare: Cloud Process Support for Opioid Recovery Participation and Learning
Brief Title: Reward-Based Recovery Outcomes Management for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Decision Logic, Inc. (Industry)
Collaborators: PRO Health Group (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-001; 1R43DA051298-01A1 (NIH)
Record Dates: First submitted 2020-11-19; First posted 2020-12-16 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROCare (Experimental): Technology-enabled, reward-based recovery platform
  Interventions: Behavioral: PROCare
- Control (No Intervention): Treatment-as-Usual

INTERVENTIONS:
Behavioral: PROCare — PROCare is a reward-based digital recovery management platform for individuals receiving medication treatment for opioid use disorder. Patients have the opportunity to earn both non-monetary and monetary incentives via smart debit card for a variety of clinically-indicated behaviors, including taking their medication (buprenorphine) as directed, attending clinic appointments and community-based mutual-help support group meetings, participating in routine outcomes monitoring surveys using validated measures, accessing the curated psychoeducation content library, and engaging in other recovery-oriented activities within the smartphone app.
  Arms: PROCare

SUMMARY:
A randomized pilot study assessing feasibility, acceptability, and preliminary effectiveness of a reward-based recovery management platform (PROCare) designed to enhance participation in outcomes monitoring, engagement in treatment care, and adherence to medication for opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* access to internet-enabled smartphone device
* primary DSM-5 opioid use disorder diagnosis
* receiving medication treatment for opioid use disorder with buprenorphine
* English language proficient

Exclusion Criteria:

* active suicidal ideation or psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Proctor, PhD, Principal Investigator — PRO Health Group; Allen Tien, MD, Principal Investigator — Medical Decision Logic, Inc.
Locations (1):
- South Florida Behavioral Health Network, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PROCare Recovery: PROCare Recovery is a technology-enabled, reward-based digital recovery management mobile app for individuals receiving medication treatment for opioid use disorder. Patients have the opportunity to earn both non-monetary and monetary incentives via smart debit card for a variety of clinically-indicated behaviors, including taking their medication (buprenorphine) as directed, attending clinic appointments (e.g., therapy sessions) and community-based mutual-help support group meetings, participating in routine outcomes monitoring surveys using validated measures, accessing the curated psychoeducation content library, and engaging in other recovery-oriented activities within the app.
Period: Overall Study
Arm/Group | PROCare Recovery | Control
Started | 8 | 5
Completed | 7 | 4
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- PROCare Recovery: Technology-enabled, reward-based recovery mobile app
- Total: Total of all reporting groups
Arm/Group | PROCare Recovery | Control | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.00 (10.76) | 33.80 (4.55) | 36.38 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Fully-Adherent to Buprenorphine
Description: Assessed by % of participants fully-adherent to daily doses during study period with higher values indicating greater buprenorphine adherence.
Time Frame: 4-week
Measure: Count of Participants; unit: Participants
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
Participants | 6 | 3

2. Primary Outcome: Percentage of Participants Fully-Adherent to Care Plan
Description: Assessed by % of participants fully-adherent to weekly outpatient individual therapy visits, community-based mutual-help recovery support meetings, and other scheduled appointments attended during study period with higher values indicating greater care plan adherence.
Time Frame: 4-week
Measure: Count of Participants; unit: Participants
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
Participants
  All Appointments | 4 | 2
  Therapy Sessions | 6 | 3

3. Primary Outcome: Percentage of Participants Completing Outcomes Monitoring Surveys
Description: Assessed by % of participants completing assessment surveys during study period with higher values indicating greater survey participation.
Time Frame: 4-week
Measure: Count of Participants; unit: Participants
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 8 | 5
Participants | 7 | 4

4. Secondary Outcome: Percentage of Participants Using Opioids
Description: Assessed by participant self-report and positive urine drug screens completed at routine clinic visits during study period.
Time Frame: 4-week
Measure: Count of Participants; unit: Participants
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
Participants | 1 | 1

5. Secondary Outcome: Percentage of Participants Using Other Substances (Non-opioids)
Description: Assessed by participant self-report and positive urine drug screens completed at routine clinic visits during study period for non-opioids substances (alcohol, cannabis, methamphetamine, amphetamines, cocaine, benzodiazepines).
Time Frame: 4-week
Measure: Count of Participants; unit: Participants
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
Participants | 2 | 2

6. Secondary Outcome: Change in Quality of Life as Assessed by EUROHIS-QOL 8-item Index From Baseline to 4-Week Follow-up
Description: The EUROHIS-QOL (European Health Interview Survey-Quality of Life) 8-item index is an efficient, valid, and reliable measure of four quality of life domains (physical, psychological, environmental, and social). Items are rated on a 5-point Likert-type scale and summed to produce a total quality of life score (Range: 8-40) with higher scores indicating a higher level of satisfaction with their current quality of life. Change in scores from baseline to 4-week follow-up was examined with a higher change score indicating a greater increase in participant quality of life.
Time Frame: 4-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
score on a scale | 4.57 (7.09) | 1.50 (9.88)

7. Secondary Outcome: Change in Opioid Craving as Assessed by Opioid Craving Scale (OCS) From Baseline to 4-Week Follow-up
Description: OCS is a 3-item measure of opioid craving with acceptable internal consistency, reliability, and concurrent/predictive validity. Participants rate their level of craving in reference to three situations (current, past week, and high-risk environment) on a scale ranging from 0-10 to produce a total score ranging from 0-30 with higher scores indicating greater reduction in craving. Change in OCS scores from baseline to 4-week follow-up was examined to determine reductions in craving.
Time Frame: 4-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
score on a scale | 19.42 (22.69) | 16.50 (22.13)

8. Secondary Outcome: Motivation as Assessed by Readiness Ruler
Description: Readiness Ruler is a valid and reliable 2-item measure of motivation and readiness to change. Participants rate their perceived "Importance" of making a change to their drug use behaviors, and their perceived "Confidence" in their ability to successfully achieve their goal (range: 0-100) with higher scores indicating greater motivation. Perceived "Importance" and "Confidence" scores are averaged to indicate a total Motivation score at 4-week follow-up (Range: 0-100).
Time Frame: 4-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
score on a scale | 93.49 (6.45) | 89.31 (13.69)

9. Secondary Outcome: Change in Self-Efficacy as Assessed by Brief Situational Confidence Questionnaire (BSCQ) From Baseline to 4-Week Follow-up
Description: BSCQ is an 8-item measure of self-efficacy for resisting the urge to use drugs in 8 high-risk situations based on the relapse prevention model (unpleasant emotions, physical discomfort, pleasant emotions, testing control, urges/temptations, interpersonal conflict, social pressure, and pleasant times with others). Patients rate their confidence in resisting the urge to use drugs in each of the 8 situations on a scale ranging from 0 (Not at all Confident) to 100 (Extremely Confident). Scores for each of the 8 situations are averaged to produce a total self-efficacy score (Range: 0-100). Change in scores from baseline to 4-week follow-up was examined with higher scores indicating a greater increase in self-efficacy.
Time Frame: 4-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
score on a scale | 54.62 (16.18) | 38.44 (25.52)

10. Secondary Outcome: Change in Opioid Use Disorder Impairment From Baseline to 4-Week Follow-up
Description: Participant self-report will be used to determine frequency counts of the 11 opioid use disorder diagnostic criteria per Diagnostic & Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) with higher counts indicating a greater number of symptoms/opioid-related impairment present and higher opioid use disorder severity. Total score indicating the total number of positive diagnostic criteria ranges from 0-11. Change in the number of diagnostic criteria endorsed from baseline to 4-week follow-up was examined to determine reduction in opioid-related impairment with higher scores indicating a greater reduction in symptoms over time.
Time Frame: 4-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 4
score on a scale | 9.86 (1.86) | 7.50 (5.74)

11. Other Pre Specified Outcome: Usability of PROCare App as Assessed by System Usability Scale (SUS)
Description: SUS is a 10-item measure commonly used for global assessments of systems usability. SUS scores will be used to objectively quantify the usability of the PROCare recovery app. Participants allocated to the PROCare condition will rate the usability of the app on 10 items assessing different aspects of usability using a Likert-type scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) with higher converted total scores indicating a higher level of overall usability. Converted total scores range from 0-100 with SUS scores above 68 considered Above Average.
Time Frame: 4-week
Population: Only participants who used the PROCare Recovery app were administered the measure of app usability.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROCare Recovery: Technology-enabled, reward-based recovery platform
  PROCare Recovery is a reward-based digital recovery management platform for individuals receiving medication treatment for opioid use disorder. Patients have the opportunity to earn both non-monetary and monetary incentives via smart debit card for a variety of clinically-indicated behaviors, including taking their medication (buprenorphine) as directed, attending clinic appointments and community-based mutual-help support group meetings, participating in routine outcomes monitoring surveys using validated measures, accessing the curated psychoeducation content library, and engaging in other recovery-oriented activities within the app.
Arm/Group | PROCare Recovery | Control
Number analyzed (Participants) | 7 | 0
score on a scale | 88.93 (10.49) |

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | PROCare Recovery | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

LIMITATIONS AND CAVEATS:
Recruitment challenges due to COVID-19 pandemic (lower patient volumes/admissions, funding, staff shortages) leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04669249/Prot_SAP_000.pdf